CLINICAL TRIAL: NCT05421962
Title: Ketamine as the Main Analgesic Agent During Analgesia-based Sedation for Elective Colonoscopy- a Randomised, Double-blind, Control Study
Brief Title: Analgosedation for Elective Colonoscopy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Mirza Kovacevic, Principal Investigator, Cantonal Hospital Zenica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMA
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pain; Side Effect
Keywords: analgesic; ketamine; fentanyl; colonoscopy
MeSH Terms: conditions — Pain | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midazolam and Fentanyl (Experimental): Patients were premedicated with 0.05 mg kg-1 of midazolam (PanPharma), 5 minutes before the starting of the procedure. Afterwards, sedation induction was performed with 1 mcg kg-1 of fentanyl (Panpharma; SanMed) and 0.5 mg kg-1 of propofol (Fresenius Kabi; Amicus Pharma).
  Interventions: Drug: Ketamine
- Midazolam and Ketamine (Experimental): Patients were premedicated with 0.05 mg kg-1 of midazolam (PanPharma), 5 minutes before the starting of the procedure. Afterwards, sedation induction was performed with ketamine (Inresa Arzneimittel) 0.5 mg kg-1 and 0.5 mg kg-1 of propofol.
  Interventions: Drug: Ketamine
- Midazolam and Propofol (No Intervention): Patients were premedicated with 0.05 mg kg-1 of midazolam (PanPharma), 5 minutes before the starting of the procedure. Afterwards, sedation induction was performed with 1 mg kg-1 of propofol.

INTERVENTIONS:
Drug: Ketamine — Ninety patients were included and randomized to either fentanyl-propofol (Group FP, n: 30), ketamine-propofol (Group KP, n: 30) or propofol-control group (Group C, n: 30). Group FP patients received fentanyl and propofol, Group KP received ketamine and propofol and Group C, propofol.
  Other Names: Fentanyl
  Arms: Midazolam and Fentanyl; Midazolam and Ketamine

SUMMARY:
Aim: The aim of the study was to to compare the analgesic effects of ketamine over fentanyl combined with propofol in analgesia-based elective colonoscopy with purpose of patient safety and satisfaction.

Methods: This is a double-blinded prospective randomized controlled trial. Ninety patients were included and randomized to either fentanyl-propofol (Group FP, n: 30), ketamine-propofol (Group KP, n: 30) or propofol-control group (Group C, n: 30). Group FP patients received fentanyl and propofol, Group KP received ketamine and propofol and Group C, propofol. In all groups, incremental doses of propofol were used to maintain a Ramsay sedation score (RSS) of 5. Respiratory depression, hemodynamic parameters were monitored for the first minute and every 5 minutes during endoscopy. Fifteen minutes after the procedure, the degree of pain was assessed using a visual analog scale (VAS), the quality of recovery according to the Aldrete score (ARS), complications during and after the procedure and additional doses of propofol were recorded.

DETAILED DESCRIPTION:
This prospective, randomized control study was conducted after obtaining the approval of the Ethics Committee and the written consent of the patients, in the Department of Anesthesia and Intensive care unit between 2020 and 2021. Ninety ASA physical statuses I and II, patients who were older than 18 years were included in this study. Exclusion criteria were: all colonoscopies lasting longer than 30 minutes, patients with previous abdominal surgery, patients treated for neuropathic pain, malignant and respiratory diseases, pregnant women, gastrointestinal obstruction, patients using antihypertensive and antiarrhythmic drugs, psychiatric patients, patients with ASA physical status III and higher, and patients who refused to participate in the study.

All patients had fasted for the previous 8 hours prior to the procedure and had undergone a digestive tract preparation procedure. Patients were randomly (computer generated) divided into three groups: patients whom were administrated fentanyl and propofol (Group FP), patients whom were administrated ketamine and propofol (Group KP) and patients whom were administrated propofol (Group C-control group). The syringes were coded before the procedure by an anesthetist who was not involved in the sedation process. Syringes were also selected in terms of volume in a similar manner, while patients, anesthesiologists, colonoscopists, and anesthetists were blinded to the medication regimen.

After the patient admission to the endoscopy room and identification, an intravenous line was placed and intravenous fluid administration (saline) was started. All patients were placed in the lateral position and placed on non-invasive blood pressure monitoring, three-channel ECG and peripheral oxygen saturation. Oxygen support is provided via a facial mask at a flow rate of 5 L/min.

Sedation protocol. All three groups of patients were premedicated with 0.05 mg kg-1 of midazolam (PanPharma), 5 minutes before the starting of the procedure. Afterwards, sedation induction was performed with 1 mcg kg-1 of fentanyl (Panpharma; SanMed) and 0.5 mg kg-1 of propofol (Fresenius Kabi; Amicus Pharma) for Group FP. Ketamine (Inresa Arzneimittel) 0.5 mg kg-1 and 0.5 mg kg-1 of propofol for Group KP, and 1 mg kg-1 of propofol for Group C. During the procedure, the patients RSS scores was maintained at 5 with an additional 0.5 mg kg-1 bolus dose of propofol when required.

Data collection and measurements Assessment of hemodynamic and respiratory stability. MAP and HR were noted upon entry of the patient into the endoscopic cabinet, immediately after the administration of propofol, and then every 5 minutes during the procedure. A number of episodes of hypertension, hypotension, tachycardia, and bradycardia were noted. Hypertension is defined as an increase in blood pressure greater than 20%, and hypotension for a decrease in blood pressure greater than 20% from baseline. Tachycardia is defined as an increase in heart rate> 100 beats per minute. Bradycardia as a drop in heart rate <50 beats per minute. Respiratory stability was assessed at the same time intervals using a peripheral pulse oximeter. A number of desaturation episodes were recorded for each group. Desaturation was defined as a decrease in peripheral oxygen saturation <95% measured with a pulse oximeter.

Assessment of sedation level. The degree of sedation were assessed by RSS, immediately after propofol administration and every 5 minutes during the procedure. RSS is a subjective method of sedation assessment, where patient sedation levels are divided into 6 groups (1. anxious, agitated or anxious or both; 2. cooperative, oriented and calm; 3. calm, responds only to command; 4. quick response to audible stimulus or light tapping on the forehead; 5. slow response to sound stimulus or light tapping on the forehead; 6. no response to stimulus). A number of additional bolus doses were recorded for each group.

Assessment of postprocedural abdominal pain. The patient's subjective feeling of post-procedural pain were determined by a 10 cm VAS. The scale is horizontal, ungraded, bounded at both ends by vertical lines that define the extreme limits of the indicators being measured. The experienced pain sensation were marked by the patient on a scale, and then the marked position were assigned a numerical value according to the VAS score as follows: VAS score: no pain 0-10 mm; mild pain 10-30 mm; moderate pain 30-70 mm; severe pain 70-100 mm. Assessment of postprocedural pain were performed 15 minutes after the procedure.

Recovery quality assessment. The quality of the patient's recovery were assessed by ARS 15 minutes after the end of the procedure. Using ARS we examined the following five criteria: motor activity (possibility of moving 2 extremities/all extremities, no movement of extremities on command), breathing (deep breathing with cough reflex, hypoventilation, apnea), blood pressure (+20 mmHg, + 20-50 mmHg, +50 mmHg relative to baseline), consciousness (awake, awake on call, unresponsive) and skin color (pink, pale, cyanotic). With ARS, each criterion is evaluated separately from 0 to 2, with a maximum score of 10. A score with a range of 8 and 9 is considered satisfactory.

Estimation of complication frequency. The frequency of procedural complications was monitored: hallucinations, confusion, unpleasant dreams, anxiety, weakness, vomiting and nausea. Hallucinations were defined as a visual or auditory sensory event that occurs without appropriate objective sensory stimulation. Confusion were defined as an inability to think clearly, an expression of a disorder of consciousness, and unpleasant dreams as an unpleasant mental activity during sleep. Anxiety were defined as a feeling of general tension, anxiety, great stress, panic or fear, and weakness as a feeling of loss of muscle strength, general fatigue or functional limitation. Vomiting were defined as a reflex act, during which the contents of the stomach or the initial part of the small intestine return through the mouth and are expelled into the external environment. Nausea were defined as a feeling of discomfort in the upper part of the digestive system with a feeling of threatening vomiting. Patients were interviewed to mark the experienced feeling with YES or NO.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical statuses I and II,
* patients who were older than 18 years

Exclusion Criteria:

* colonoscopies lasting longer than 30 minutes,
* patients with previous abdominal surgery,
* patients treated for neuropathic pain, malignant and respiratory diseases,
* pregnant women, gastrointestinal obstruction,
* patients using antihypertensive and antiarrhythmic drugs,
* psychiatric patients,
* patients with ASA physical status III and higher,
* patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Degree of the pain | 15 minutes
  15 minutes after the procedure, the degree of pain was assessed using a visual analog scale (VAS).The scale is horizontal, ungraded, bounded at both ends by vertical lines that define the extreme limits of the indicators being measured. The experienced pain sensation were marked by the patient on a scale, and then the marked position were assigned a numerical value according to the VAS score as follows: VAS score: no pain 0-10 mm; mild pain 10-30 mm; moderate pain 30-70 mm; severe pain 70-100 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital, Zenica, Bosnia and Herzegovina